CLINICAL TRIAL: NCT05900739
Title: Social Media for Nutrition Education. Fruit and Vegetable Intake Promotion in a University Setting: "The UVa Community Eats Healthy" Study Protocol
Brief Title: Fruit and Vegetable Intake Promotion. "The UVa Community Eats Healthy" Study Protocol (University of Valladolid)
Acronym: UVa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Laura Carreño Enciso, Associated Professor, University of Valladolid
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13022022
Record Dates: First submitted 2023-04-20; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Fruit and Vegetable Consumption

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1: Virtual Campus (Experimental): This group received 7 sessions (one every 7 days) of one hour through moodle virtual campus (webinar) to work TPB constructs: attitude; subjective norms; perceived behavioural control and intention.
  Interventions: Behavioral: Increase of fruit and vegetable consumption
- Intervention 2: Facebook (Experimental): This group received 25 educational impacts (2-5 per week - during 7 weeks) through a private group of facebook. Activities were: posts, stories and Facebook Lives as workshops (recorded)
  Interventions: Behavioral: Increase of fruit and vegetable consumption
- Intervention 3: Instagram (Experimental): This group received 35 educational impacts (4-6 per week - during 7 weeks) through a private account of instagram. Activities were: posts, stories and Instagram Lives as workshops (recorded)
  Interventions: Behavioral: Increase of fruit and vegetable consumption
- Control (No Intervention): Information about Mediterranean Diet was provided but no activities nor interventions took place.

INTERVENTIONS:
Behavioral: Increase of fruit and vegetable consumption — Week 1 Presentation of the program. Healthy eating Week 2 Fruit and vegetable: nutritional value, types, seasonality, benefits for health Week 3 Shopping Fruit and vegetable: tips, places, conservation methods Week 4 Healthy menu planning with "My Plate" Week 5 How to cook Fruit and Vegetable avoiding food waste Week 6 Healthy snacks using Fruit and vegetable Week 7 Batch cooking
  Arms: Intervention 1: Virtual Campus; Intervention 2: Facebook; Intervention 3: Instagram

SUMMARY:
The goal of this randomized controlled trial is to increase the consumption of fruit and vegetables of the University of Valladolid (UVa) community employing three different online methodologies: facebook (FB), virtual campus (VC) and, instagram (IG).

DETAILED DESCRIPTION:
In order to use different methodologies, the sample was randomly divided in four groups, three took the nutrition educational program and the other one was a control group.

All four groups had access to the virtual campus of the UVa which uses the teaching platform Moodle Learning Management System (LMS). In this platform, a course entitled "The UVa community eats healthy" was created with four sections. Each of the sections corresponded to one of the four groups, the names of the sections were: I-campus (VC group), C-campus (control group), F-campus (FB group), and G-campus (IG group).

To make the intervention more effective, this program was theory-based designed, based on the theory of planned behaviour (TPB).

In order to assess the effectivity of social media use for nutrition education compared to more traditional interventions, the program was adapted to three platforms: virtual campus, private account of IG and private group of FB. The topics of the intervention groups were the same but with adapted activities.

ELIGIBILITY:
Inclusion Criteria:

* being part of the UVa community at the time of recruitment
* having IG and/or FB account
* having made the self-registration to the Moodle virtual campus of each group during the enrolment period

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable consumption | up to 8 weeks
  The consumption will be measured using MEDAS-14 questionnaire from Predimed Study

SECONDARY OUTCOMES:
Fruit and vegetable consumption of the different groups | up to 8 weeks
  The consumption will be measured using MEDAS-14 questionnaire from Predimed Study classified by group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No